CLINICAL TRIAL: NCT06458036
Title: Selpercatinib to Enhance RAI Avidity in Children, Adolescents, and Young Adults With Newly Diagnosed Differentiated Thyroid Cancers Harboring RET Fusions
Brief Title: Selpercatinib Pre-RAI in Patients With RET Fusion Thyroid Cancer (RAISE)
Acronym: RAISE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Eli Lilly and Company (Industry); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-021524
Record Dates: First submitted 2024-06-10; First posted 2024-06-13 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Differentiated Thyroid Cancer; Pediatric Cancer; Cancer; Cancer, Thyroid
Keywords: Thyroid Cancer
MeSH Terms: conditions — Neoplasms; Thyroid Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: Selpercatinib Monotherapy with 131I Therapy (Experimental): Patients will receive selpercatinib monotherapy for 6 months at the FDA-approved dose.
  Patients will receive 131I therapy after 6 months of selpercatinib. Selpercatinib will be continued for 5 days after RAI therapy and then patients will enter a wait and see period off treatment.
  Patients who experience disease progression at any point while on selpercatinib will proceed to 131I therapy and discontinue selpercatinib.
  Interventions: Drug: Selpercatinib Monotherapy; Radiation: 131I Therapy

INTERVENTIONS:
Drug: Selpercatinib Monotherapy — Patients will receive selpercatinib monotherapy for 6 months at the FDA-approved dose.
Radiation: 131I Therapy — Patients will receive 131I therapy after 6 months of selpercatinib.

SUMMARY:
Papillary thyroid cancer (PTC) is the most common form of differentiated thyroid cancer (DTC). The traditional first line treatment for patients with advanced DTC after surgical resection is radioactive iodine (RAI) therapy. However, less than a quarter of patients with lung metastases will achieve a complete response to RAI therapy, and this therapy carries the risk of pulmonary fibrosis and an increasingly recognized risk of secondary malignancies.

DETAILED DESCRIPTION:
This will be an open label, non-randomized study to evaluate the efficacy and safety of the combination of selpercatinib followed by 131I therapy for patients with RET fusion differentiated thyroid cancer. The primary Phase II objective will be to evaluate the pulmonary structural response rate at 18 months to the combination of selpercatinib given for 6-months followed by 131I therapy. This is exempt from Investigational New Drug requirements per the FDA.

ELIGIBILITY:
Inclusion Criteria:

1. Age 2-25 years, inclusive
2. Histologic diagnosis of a differentiated thyroid cancer, status post thyroidectomy and adequate local therapy (e.g., lymph node dissection as per standard of care) for metastatic disease in the neck in the opinion of the treating investigator
3. Anatomically evaluable disease on chest CT (Computed Tomography) meeting one of the following criteria (obtained within 90 days of enrollment):

   A. multiple (> 10) noncalcified solid pulmonary nodules visible on CT and/or B. enlarging, discrete pulmonary nodules visible on CT of any number consistent with metastatic disease
4. Identification of an activating RET gene alteration (fusion or mutation). The RET alteration result should be generated from a laboratory with specific certifications (depending on country requirement) that clearly denotes the presence of a RET alteration without known kinase domain resistance mutation
5. Lansky/Karnofsky performance status >50%
6. Adequate Organ Function

   A. Bone Marrow Function:
   * Peripheral absolute neutrophil count (ANC) ≥1500/µL
   * Platelet count ≥ 100,000/µL (transfusion independent, defined as not receiving platelet transfusions for at least 7 days prior to enrollment)
   * Hemoglobin ≥ 9.0 g/dL at baseline (may receive Red Blood Cell transfusions).

   B. Adequate Renal Function: Creatinine clearance or radioisotope Glomerular Filtration Rate (GFR) ≥ 70 mL/min/1.73 m2 or a maximum serum creatinine based on age/gender.

   C. Adequate Liver Function
   * Bilirubin (sum of conjugated + unconjugated) < / = 1.5 x upper limit of normal (ULN) for age. Except participants with a documented history of Gilbert syndrome who must have a total bilirubin level of <3.0X ULN
   * Alanine aminotransferase (ALT) <2.5X ULN OR <5x ULN if the liver has tumor involvement. For the purpose of this study, the ULN for ALT is 45 U/L.
   * Serum albumin ≥ 2 g/dL
7. Patient must have normal serum potassium, calcium, and magnesium levels (may be receiving supplements)
8. Men with partners of childbearing potential or women of childbearing potential must agree to use a highly effective contraceptive method during treatment with study drug and for 6 months following the last dose of study drug. Selpercatinib could impair fertility in males and females. Advise women not to breastfeed during treatment with selpercatinib and for 1 week following the final dose
9. Women of childbearing potential must have a negative pregnancy test (serum or urine, consistent with local regulations) documented within 24 hours prior to treatment with study drug and at least monthly while on study treatment

Exclusion Criteria:

1. No prior systemic therapy for thyroid cancer, including RET inhibitors. Note: prior 131I is allowed.
2. Females who are pregnant or breastfeeding are excluded due to the potential risks of selpercatinib and radioactive iodine to the fetus/neonate.
3. Concurrent therapy: Patients currently receiving a strong CYP3A4 inducer or inhibitor are not eligible. Strong inducers or inhibitors of CYP3A4 should be avoided 14 days prior to treatment to the end of the study treatment.
4. Patients with clinically significant active cardiovascular disease, Torsades de pointes, or history of myocardial infarction within 6 months prior to planned start of study treatment or prolongation of the QT interval corrected for heart rate using Fridericia's formula (QTcF) >470 msec.
5. Have clinically significant active malabsorption syndrome or other condition likely to affect gastrointestinal absorption of the drug.
6. Are taking a concomitant medication that is known to cause QTc prolongation.
7. Active hemorrhage or at significant risk for hemorrhage.
8. Uncontrolled hypertension (blood pressure greater than 140/90 in adults or greater than the 95% for height and gender in children). Use of anti-hypertensives to control blood pressure is permitted.

Ages: 2 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-07-29 (Actual); Primary Completion 2030-11-01 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of patients with complete overall, pulmonary, structural, and biochemical response. | 18 months
  Determine the overall, pulmonary, structural, and biochemical response rate to selpercatinib in patients with RET fusion differentiated thyroid cancer treated with 6 months of selpercatinib prior to 131I therapy
Number of patients who survive without progression of disease after 5 years following protocol treatment. | 5 years
  Determine the progression free survival to the combination of selpercatinib followed 6 months later 131I therapy from the initiation of selpercatinib therapy
Proportion of all patients enrolled who show increased radioactive iodine avidity at 6 months following selpercatinib monotherapy. | 6 months
  Determine the proportion of patients for whom oncogene-specific, targeted therapy increases tumor RAI-avidity.
The incidence of adverse events and dose limiting toxicity with the combination of selpercatinib and 131I therapy, graded according to CTCAE v5. | 12 months
  Determine the safety of the combination of selpercatinib given for 6-months followed by 131I therapy in patients with RET fusion differentiated thyroid cancer

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Laetsch, MD, Principal Investigator — Children's Hospital of Philadelphia
Locations (2):
- United States (2):
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Hospital, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No